CLINICAL TRIAL: NCT03598179
Title: A Single-center, Open Study Evaluating Efficacy and Safety of XLCART001（CD-19） Treatment in Relapsed/Refractory/High-risk B-cell Malignancy Subjects
Brief Title: XLCART001 Treatment in Relapsed/Refractory/High-risk B-cell Malignancy Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, JianYong Li, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-CART001
Record Dates: First submitted 2018-06-27; First posted 2018-07-26 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma, B-Cell; Leukemia, B-cell
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: chimeric antigen receptor T cells — Dose CAR+ cells/kg B-cell lymphoma 4×10^6 Acute lymphocytic leukemia 2×10^6 Chronic lymphocytic leukemia 10×10^6

SUMMARY:
The trial is a single arm, single-center, non-randomized clinical trial which is designed to evaluate the efficacy and safety of XLCART001 in treatment of relapsed/refractory/high-risk B-cell malignancy subjects

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male and female,
* Confirmed as CD19-positive B cell lymphoma/leukemia by immunohistochemistry or flow cytometry
* No effective treatment
* Patients must have a measurable or evaluable disease at the time of enrollment.
* Adequate organ system function including:

  * ALT/AST < 3 upper limit of normal; Total Bilirubin < 2.5 upper limit of normal
  * Creatinine < 2 upper limit of normal
  * Oxygen saturation ≥ 95%
  * Left ventricular ejection fraction ≥ 40%
  * Number of neutrophil ≥ 0.75×10^9/L, number of platelet ≥ 50×10^9/L
* At least 4 weeks from receiving previous treatment (radiotherapy, chemotherapy, monoclonal antibody therapy or other treatments)
* No contraindications of peripheral blood apheresis
* Female subjects in childbearing age, their serum or urine pregnancy test must be negative. All patients must agree to take effective contraceptive measures during the trial measures
* ECOG score 0-2, expected survival ≥ 12 weeks

Exclusion Criteria:

* Women who are pregnant or lactating. Patients have breeding intent in 12 months or cannot take effective contraceptive measures during the trial measures
* Uncontrollable active infection within four week. Prophylactic antibiotic, antiviral and antifungal treatment is permissible. Active hepatitis B or hepatitis C virus infection, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV-infected persons
* Subjects with any autoimmune disease or any immune deficiency disease
* Have a history of allergy to antibodies or cellular products
* Participated in any other clinical trial within four weeks
* Used of systemic steroids within four weeks (using inhaled steroids or ≤ 20mg/d prednison are exceptions)
* Have mental diseases
* Have history of drug addiction
* The investigators believe that any increase in the risk of the subject or interference with the results of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 12 weeks
  Overall response rate (ORR) = complete response (CR) rate + partial response (PR) rate, ORR will be assessed at weeks 12.
Overall Survival | 6 months,1 year, 2 years
  from the time of enrollment to death from any cause or the date of the last follow-up visit
Progression-free Survival | 12 weeks,6 months,1 year, 2 years
  the time from enrollment to disease progression, death from any cause, or the date of the last follow-up visit
Event-free Survival | 12 weeks,6 months,1 year, 2 years
  the time from enrollment to any events, or the date of the last follow-up visit

SECONDARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
  Non-haematological dose-limiting toxicities was any toxicity of grade 3 or higher occurring within 28 days of XLCART001 infusion judged possibly related to the treatment regimen.The following toxicities were not considered dose limiting toxicities: tumor lysis syndrome, abnormal electrolytes responding to supplementation, hypoalbuminemia, liver dysfunction resolving to ≤grade 2 within 14 days, transient (<72 hours) grade 4 hepatic enzyme abnormality, and grade 3 or 4 fever or neutropenic fever.
Number of CAR-T cells | Day 1, Day 4, Day 7, Day 10, Day 14, Day 21, Day 28, 8 weeks, 12 weeks, 6 months, 1 years, 2 years
  The number of CAR-T cells detected by flow cytometry and copy number of CAR-T cells tested by polymerase chain reaction
Duration of CAR-T cells | Day 1, Day 4, Day 7, Day 10, Day 14, Day 21, Day 28, 8 weeks, 12 weeks, 6 months, 1 years, 2 years
  The duration of CAR-T cells detected by flow cytometry and copy number of CAR-T cells tested by polymerase chain reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Haematology, the First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjin, Jiangsu, China

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338